CLINICAL TRIAL: NCT03531736
Title: Allogeneic Hematopoietic Stem Cell Transplantation of α/β T-Lymphocyte Depleted Graft Conditioned With a Reduced Intensity Regimen in Patients With Hematologic Malignancies and Aplastic Anemia
Brief Title: T Cell Depleted Allogeneic Hematopoietic Stem Cell Transplantation Conditioned With a Reduced Intensity Regimen in Patients With Hematologic Malignancies and Aplastic Anemia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-639
Record Dates: First submitted 2018-05-09; First posted 2018-05-22 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Myeloid Diseases
Keywords: Allogeneic Hematopoietic Stem Cell Transplantation; intensity conditioning regimen; 17-639
MeSH Terms: interventions — thymoglobulin; fludarabine; Whole-Body Irradiation; Cyclophosphamide; Rituximab

STUDY DESIGN:
Intervention Model Description: This is a pilot study to assess engraftment of a T cell depleted (TCD) graft following a reduced intensity conditioning regimen (RIC). The conditioning regimen will include total body irradiation (TBI), Fludarabine, anti-thymocyte globulin (ATG) and post transplant cyclophosphamide (PT-Cy). The graft will be TCD and will be composed of a TCR-α/β+ lymphocyte depletion stem cells and CD34+ selected stem cells.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients with Myeloid Malignancies & Aplastic Anemia (Experimental): Transplant conditioning will consist of: ATG (2 mg/kg/day IV on days-8 through-6), fludarabine (30 mg/m^2/d on days -5 through -2), TBI 400 cGy in 2 divided doses (days -2 and -1) and high dose cyclophosphamide given post stem cell infusion (50 mg/kg on days +3 and +4). One dose of Rituxan (200 mg/m^2) will be given to reduce the risk of EBV viremia. The donor stem cell product will be derived from the peripheral blood with a target cell infusion of ≥8X10^6 CD34 cells per recipient kg. Patients will receive post-transplant G-CSF starting on day +7. Patients will undergo donor/recipient bone marrow and peripheral chimerism studies at 30 and 100, and 6, 12, 18 and 24 months post allo HCT and thereafter, at the discretion of the treating clinician. Immune function and disease restaging will be performed at day 100 and 6, 12, 18, and 24 months and as otherwise clinically indicated by the treating physician.
  Interventions: Drug: Antithymocyte globulin (Rabbit); Drug: fludarabine; Radiation: total body irradiation; Drug: cyclophosphamide; Drug: Rituxan; Procedure: Allogeneic Hematopoietic Stem Cell Transplantation

INTERVENTIONS:
Drug: Antithymocyte globulin (Rabbit) — ATG (2 mg/kg/d IV on days-8 through -7)
  Other Names: ATG
Drug: fludarabine — fludarabine (30 mg/m2/d on days -5 through -2)
Radiation: total body irradiation — TBI 200 cGy (days -2 and -1) given post stem cell infusion
  Other Names: TBI
Drug: cyclophosphamide — cyclophosphamide given post stem cell infusion (50 mg/kg on days +3 and +4)
Drug: Rituxan — Rituxan (200 mg/m2) will be given to reduce the risk of EBV viremia
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Allogeneic Hematopoietic Stem Cell Transplantation

SUMMARY:
The main purpose of this study is to learn if a new combination of chemotherapy, in combination with low-dose radiation, will be safe for the patient, and at the same time provide the best opportunity to cure the bone marrow cancer. The combination of chemotherapy and radiation described in the study is considered 'low intensity.' Although the chemotherapy agents used in this study and for transplant are FDA approved, the chemotherapy treatment and conditioning regimens or combinations listed in this consent are not yet FDA approved.

The CliniMACS device is FDA approved for one type of T cell depletion (positive selection of the stem cells) but not approved yet for other type of T cell depletion, which is being studied on this protocol. This pilot study, along with other studies will serve as the basis for FDA approval, if outcomes are favorable.

ELIGIBILITY:
Inclusion Criteria:

* Patients with one of the high risk myeloid diseases as outlined below. Patients must have ≤ 5% blasts on the last BM evaluation prior to starting the conditioning regimen. Diseases included on this protocol include:

  1. Acute Myeloid Leukemia (AML) in CR1 with intermediate or high risk features as defined below:

     °Cytogenetic abnormalities which are not considered "good risk" cytogenetic features (i.e t(8:21), t(15:17), inv 16 without c-kit mutations.

     And/or
     * Therapy related AML with history of antineoplastic therapy (radiation and/or chemotherapy) And/or
     * Normal karyotype with mutations of FLT3, RUNX1, TP53 mutation, ASXL1 or any others that are considered to be high risk
  2. AML in ≥ 2nd remission
  3. Myelodysplastic syndrome, myeloproliferative neoplasms, or MDS/MPN overlap syndrome with:

     °International prognostic scoring system risk score INT-2 or high risk at the time of transplant evaluation.

     And/or
     * Any risk category if life-threatening cytopenia exists And/or
     * Karyotype or genomic changes that indicate high risk for progression to acute myelogenous leukemia, including abnormalities of chromosome 7 or 3, mutations of TP53, or complex or monosomal karyotype.
  4. Chronic myelomonocytic leukemia (CMML)
  5. Chronic myeloid leukemia (CML) with the following features:

     °Patients who have failed or are intolerant to BCR-ABL tyrosine kinase inhibitors.

     And/or

     °CML with BCR-ABL mutation consistent with poor response to tyrosine kinase inhibition (e.g T351l mutation)
  6. Patients with severe aplastic anemia
* Chronic lymphocytic leukemia (CLL) with high risk disease as defined by the EBMT consensus criteria.
* Non-Hodgkin lymphoma meeting both of the following criteria:

  * Responding to therapy prior to enrollment.
  * Relapse after prior autologous bone marrow transplant or are ineligible for autologous bone marrow transplant.
* Multiple Myeloma with disease in the following categories:

  * Patients with relapsed multiple myeloma following autologous stem cell transplantation who have achieved at least partial response following additional chemotherapy
  * Patients with high risk cytogenetics at diagnosis must have achieved at least a partial response following autologous stem cell transplantation. Patients must have complex karyotype, del17p, t4;14, and/or t14;16 by FISH and/or del13 by karyotyping.
* Each patient must be willing to participate as a research participant and must sign an informed consent form.
* Organ Function and Performance Status Criteria:

  1. Patients be ≥ 18 years old.
  2. Patients must have a Karnofsky (adult) or Performance Status ≥ 70%.
  3. Patients must have adequate organ function measured by:

     * Cardiac: asymptomatic or if symptomatic, then LVEF at rest must be ≥ 40% and must improve with exercise.
     * Hepatic: < 5x ULN ALT and < 2x ULN total serum bilirubin, unless there is congenital benign hyperbilirubinemia.
     * Renal: CrCl >30ml/min (measured or calculated/estimated).
     * Pulmonary: asymptomatic or if symptomatic, DLCO > 50% of predicted (corrected for hemoglobin)

Exclusion Criteria:

* Prior allogenic hematopoietic stem cell transplantation
* Prior radiation therapy with 400cGY or more of TBI
* BM with increased fibrosis (Reticulin stain > 1/3)
* Active and uncontrolled infection at time of transplantation
* HIV infection
* Seropositivity for HTLV-1
* Inadequate performance status/ organ function
* Pregnancy or breast feeding
* Patient or guardian unable to give informed consent or unable to comply with the treatment protocol including appropriate supportive care, follow-up, and research tests.

Donor Inclusion and Exclusion Criteria:

* Must be a 10/10 HLA genotypically match related or unrelated donor at all A, B, C, DRB1, and DQB1 loci, as tested by DNA analysis
* Able to provide informed consent for the donation process per institutional standards
* Meet standard criteria for donor collection as defined by the National Marrow Donor Program Guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Rate of donor Neutrophil Engraftment | 30 days post-transplant
  Neutrophil engraftment (recovery of ANC) defined by an ANC ≥ 500/mm^3 for 3 consecutive days

CONTACTS AND LOCATIONS:
Overall Officials: Roni Tamari, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm